CLINICAL TRIAL: NCT05699837
Title: Home-based Brainwave Entrainment Technology (hBET) for Management of Chronic Pain and Sleep Disturbance: EEG Extension to a Feasibility Study
Brief Title: Alpha Entrainment for Pain and Sleep (Extension)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: University of Leeds (Other); University of Warwick (Other)
Responsible Party: Principal Investigator, Stephen Halpin, Principle investigator, University of Manchester
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: NHS001542(2)
Record Dates: First submitted 2022-11-22; First posted 2023-01-26 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Pain, Chronic; Sleep Disturbance
MeSH Terms: conditions — Chronic Pain; Parasomnias

STUDY DESIGN:
Intervention Model Description: Following a baseline period each participant will use two types of sensory stimulation for two weeks, in a randomised order, with a 1 week washout period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The stimulation is delivered via a smartphone application. Each participant will receive one of two versions, which are identical apart from the order in which the two types of stimulation are given. The participant and the investigator enrolling participants and conducting questionnaire and interview outcome assessment, will be masked as to which version they are using. The record of which version was allocated to which participant will be held centrally by co-investigators with no direct participant contact, until results are analysed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hBET 1 (Experimental): Rhythmic stimulation (2 weeks) followed by non-rhythmic stimulation (2 weeks)
  Interventions: Device: Audio or visual alpha (10Hz) stimulation
- hBET 2 (Experimental): Non-rhythmic stimulation (2 weeks) followed by rhythmic stimulation (2 weeks)
  Interventions: Device: Audio or visual alpha (10Hz) stimulation

INTERVENTIONS:
Device: Audio or visual alpha (10Hz) stimulation — Smartphone app-based brainwave entrainment programme using audio stimulation via binaural beats or visual stimulation via flickering lights, to deliver rhythmic 10Hz or non-rhythmic stimulation

SUMMARY:
Long-term pain affects one-third of the United Kingdom population and can be very disabling. People experiencing long-term pain often suffer from disturbed sleep because of their pain symptoms, and disturbed sleep can then make their pain symptoms worse. Managing long-term pain is also very costly to the National Health Service. The most common treatment is prescribed medicines, but these do not always work and can have serious side-effects for some patients.

The investigators have been developing an alternative approach for treating long-term pain. This approach uses simple non-invasive tools to promote some kinds of brain activity over others. It involves patients using headphones to listen to some specific sounds, or a headset with lights flashing at particular frequencies. The studies undertaken so far seem to show that doing this can change how the brain responds to pain. It potentially offers an inexpensive yet effective way of reducing pain and improving sleep for patients with long-term pain. There are a few small studies that support this approach and more work is needed. In a recent study the investigators found that these tools can be reliably used in home settings and there were some indications that they improved symptoms. However, sleep was only measured with sleep diary and movement detection, there was no direct measurement of whether the stimulation frequencies were resulting in the desired brainwave changes. Finally, the benefit to symptoms may have been the result of other factors, such as the passage of time or placebo effect.

Therefore this study extends the experiment, adding more accurate sleep monitoring which includes monitoring electrical activity in the brain (EEG), as well as providing rhythmic and non-rhythmic stimulation in a randomised order. The aim is to further test the effect of these home-based tools with individuals with long-term pain, in a more rigorous way. Up to 30 participants with long-term pain and pain-related sleep disturbance will use the tools for 30 minutes at bed time every day for 4 weeks (2 weeks with one type of stimulation, 2 weeks with another type). The changes in participants' pain, sleep, brainwave frequencies, fatigue and mood will be measured.

These findings will inform the planning and design of a future much larger study to test this technology, if this is justified by the results.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80 years
* Chronic non-cancer pain (recurring pain ≥ 3 months duration)
* Diagnosis of fibromyalgia, meeting 2016 ACR criteria.
* Having nocturnal pain (NRS 0-10 worst pain ≥ 4)
* Self-reported sleep difﬁculties (trouble falling asleep, difﬁculty staying asleep, waking up too early, or waking up unrefreshed) 3 or more nights per week during the past month

Exclusion Criteria:

* Planned intervention during the study period
* Seizure disorder
* Photosensitivity
* Hearing or sight problems causing inability to use hBET
* Cognitive problems or dementia or mental health disorders causing inability to consent
* Night shift worker
* Any known primary sleep disorder including obstructive sleep apnoea, narcolepsy, restless leg syndrome

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2022-09-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Change in alpha power from baseline | Daily for 6 weeks
  Alpha spectral power in active stimulation use periods compared to sham stimulation use periods relative to equivalent baseline periods.
Change in Sleep Quality from baseline, measured with Pittsburgh Sleep Quality Index | Weeks 1, 3 and 6
  Sleep quality (0-21 score) at the end of 2 week active stimulation use period compared to at the end of 2 week sham stimulation use period each relative to the baseline period.

SECONDARY OUTCOMES:
Daily pain diary | Daily for 6 weeks
  pain over 24 hours and at night (0-10 NRS)
Daily sleep diary; total sleep time | Daily for 6 weeks
  Total sleep time (minutes)
DREEM headband; total sleep time | Daily for 6 weeks
  Total sleep time (minutes)
Actigraphy; total sleep time | Daily for 6 weeks
  Total sleep time (minutes)
Daily sleep diary; sleep onset latency | Daily for 6 weeks
  Sleep onset latency (minutes)
DREEM headband; sleep onset latency | Daily for 6 weeks
  Sleep onset latency (minutes)
Actigraphy; sleep onset latency | Daily for 6 weeks
  Sleep onset latency (minutes)
Daily sleep diary; Wake after sleep onset | Daily for 6 weeks
  Wake after sleep onset (minutes)
DREEM Headband; Wake after sleep onset | Daily for 6 weeks
  Wake after sleep onset (minutes)
Actigraphy; Wake after sleep onset | Daily for 6 weeks
  Wake after sleep onset (minutes)
Daily sleep diary; Sleep Efficiency | Daily for 6 weeks
  sleep efficiency (%)
DREEM headband; Sleep Efficiency | Daily for 6 weeks
  sleep efficiency (%)
Actigraphy; Sleep Efficiency | Daily for 6 weeks
  sleep efficiency (%)
Daily sleep diary; Sleep quality | Daily for 6 weeks
  Rating of quality (0-5 NRS) and refreshed (0-5 NRS)
DREEM headband derived sleep architecture | Daily for 6 weeks
  Duration in and latency to (minutes) and proportion (%) in each stage (N1, N2, N3, REM)
DREEM headband derived microarousal index | Daily for 6 weeks
  Microarousal frequency (events/hour)
DREEM headband recorded awakenings | Daily for 6 weeks
  Awakenings (number)
Brief Pain Inventory Pain Interference score | Weekly for 6 weeks
  0-10 NRS for pain interference
Brief Pain Inventory Severity score | Weekly for 6 weeks
  0-10 NRS for pain severity
Hospital Anxiety and Depression Scale | Weeks 1, 3 and 6
  Scores of 0-21 for anxiety, 0-21 for depression
Multidimensional Fatigue Inventory | Weeks 1, 3 and 6
  Score of 20-100
EuroQol 5 Dimensions (EQ-5D-5L) | Weeks 1, 3 and 6
  0-1 global index score, 0-100 VAS score.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony KP Jones, Study Director — University of Manchester
Locations (2):
- United Kingdom (2):
  - University of Manchester, Manchester, England
  - Leeds Community Healthcare NHS Trust, Leeds

DOCUMENTS (1):
  • Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/37/NCT05699837/SAP_000.pdf